CLINICAL TRIAL: NCT06516666
Title: Psychophysiological Effects of Music on Sadness in Depressed and Non-Depressed Participants
Brief Title: Psychophysiological Effects of Music
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Shulin Chen, Professor, Zhejiang University
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Music study in China
Record Dates: First submitted 2024-07-01; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Sadness
Keywords: music; depression; emotion; heart rate variability
MeSH Terms: conditions — Depression | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depressed group (Experimental): The participants were categorized into two groups using the Patient Health Questionnaire (PHQ-9) and the 17-item Hamilton Depression Rating Scale (HAM-D). PHQ-9 is a self-report scale. PHQ-9 scores of 5 or higher represent mild and severe depression, while PHQ-9 scores of lower than 5 mean normal condition. HAM-D is a scale administered by a healthcare professional. The cut-off point of the HAM-D scale is 8, which divides normal conditions from depressive conditions. The participants first completed PHQ-9. For those with PHQ-9 scores of 5 or higher, the trained researchers interviewed them and rated their severity of depression on the HAM-D. The participants first completed PHQ-9.
  For those with PHQ-9 scores ≥ 5, the trained researchers interviewed them and rated their severity of depression on the HAM-D. Those with HAM-D scores > 8 were classified into the depressed group.
  Interventions: Behavioral: Music
- Non-depressed group (Experimental): Those with PHQ-9 scores < 5 or HAM-D scores ≤ 8 were classified into the non-depressed group.
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music — Participants went through four stages. In the rest stage, they were instructed to relax. In the neutral control stage, they watched an informative video about plastic injection molding. In the sadness induction stage, they viewed sad clips from either Hachi: A Dog's Tale or My Brother and Sister, with the order randomized across participants. In the music intervention stage, they listened to the cheerful Cuckoo Waltz. Each stage lasted for about 6 minutes.
  The interventions for the two groups were exactly same.
  PS: On the basis of the PHQ-9, this HAMD interview was conducted to further group the participants. So, following the experimental protocol, participants who scored ≥ 5 on the PHQ-9 measure underwent the HAMD interview, while the remaining individuals were simply interviewed about their feelings during the experiment.

SUMMARY:
This study employed a repeated measure between-subjects design. Two groups (i.e., depressed group and non-depressed group) of participants were recruited. Each participant experienced four stages: baseline, neutral control, sadness induction, and music intervention. The outcome variables were self-reported emotion and Heart Rate Variability features. Emotions were reported at the end of every stage. Electrocardiogram signals were recorded throughout the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years
* Right-handed
* No recent illness or medication use
* No history of neurological or psychiatric disorders
* Normal or corrected-to-normal visual acuity (myopic participants wore glasses)
* Normal hearing

Exclusion Criteria:

* Incapable of giving written informed consent to this study
* Acute high suicide risk at baseline assessment
* Psychosis

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Self-Assessment Manikin (SAM) | Immediately after the baseline, immediately after the neutral control, immediately after the sadness induction, and immediately after the music intervention.
  The SAM scale is a brief and widely used tool for assessing emotional states. The scale is a nonverbal self-report measure of emotion, using a set of cartoon-like manikins. The manikins illustrate nine intensity levels for valence (1 = unpleasant; 9 = pleasant), arousal (1 = calm, 9 = excited), and dominance (1 = controlled; 9 = controlling).
Revision of Positive Affect and Negative Affect Scale (PANAS-R) | Immediately after the baseline, immediately after the neutral control, immediately after the sadness induction, and immediately after the music intervention.
  The PANAS is another widely used scale to measure mood or emotion. The Chinese version of PANAS is comprised of 18 items, with 9 items measuring positive affect (e.g., joyful, inspired) and 9 items measuring negative affect (e.g., sad, fearful). Because participants were required to report their feelings repeatedly in this study, 18 items would be too long and tiresome. The 18 items plus "calmness" were used as 19 options for participants to choose. They needed to select one of the emotion words to tag their strongest emotion for the stage that they had just experienced. This revision of PANAS allowed us to capture the specific emotion type.
Mean of Normal-to-Normal Intervals (MeanNN) | Throughout the whole experiment, an average of 6 minutes for each stage.
  MeanNN refers to the average duration between consecutive normal heartbeats, also named inter-beat interval. A higher MeanNN indicates a lower heart rate.
Standard Deviation of Normal-to-Normal Intervals (SDNN) | Throughout the whole experiment, an average of 6 minutes for each stage.
  SDNN measures the overall variability of heart rate. Higher SDNN values indicate greater variability.

CONTACTS AND LOCATIONS:
Locations (1):
- Shulin Chen, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradley MM, Lang PJ. Measuring emotion: the Self-Assessment Manikin and the Semantic Differential. J Behav Ther Exp Psychiatry. 1994 Mar;25(1):49-59. doi: 10.1016/0005-7916(94)90063-9. PMID 7962581
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Derived] Wang X, Lu T, Zhou B, Chen W, Zheng J, Chen H, Chen S. Psychophysiological effects of music on sadness in participants with and without depressive symptoms. BMC Complement Med Ther. 2025 Feb 26;25(1):77. doi: 10.1186/s12906-025-04824-y. PMID 40011873